CLINICAL TRIAL: NCT00945828
Title: Assessing Implementation and Effectiveness of Individual Education Plans for Children With Chronic Illness
Brief Title: Assessing the Effectiveness of Individual Education Plans for Childhood Cancer Survivors
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Miami (Other)
Collaborators: American Cancer Society, Inc. (Other)
Responsible Party: Principal Investigator, Maria L. Goldman, Co-Investigator, University of Miami
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: RSGPB PBP 105184; RSGPB PBP 105184
Record Dates: First submitted 2009-07-22; First posted 2009-07-24 (Estimated); Last update posted 2012-03-08 (Estimated); Status verified 2012-03

CONDITIONS: Acute Lymphoblastic Leukemia; Central Nervous System Tumors; Lymphoma
Keywords: pediatric cancer, neurocognitive outcomes for pediatric cancer; acute lymphoblastic leukemia; central nervous system tumors; lymphoma
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma; Central Nervous System Neoplasms; Lymphoma; Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Annual Monitoring of IEP (Experimental): Parents/caregivers and the teacher of participants will be asked to evaluate the effectiveness of the child's IEP once per academic calendar year. The evaluation is done through the use of an IEP Questionnaire developed for this study.
  Interventions: Behavioral: Annual Intervention Group
- Quarterly Monitoring of IEP (Experimental): Parents/caregivers and the teacher of participants will be asked to evaluate the effectiveness of the child's IEP four times per academic calendar year. The evaluation is done through the use of an IEP Questionnaire developed for this study.
  Interventions: Behavioral: Quarterly Monitoring of IEP

INTERVENTIONS:
Behavioral: Annual Intervention Group — Parents/caregivers and the teacher of participants will be asked to evaluate the effectiveness of the child's IEP once per academic calendar year. The evaluation is done through the use of an IEP Questionnaire developed for this study. This questionnaire addresses the child's academic performance, progress, and adherence to the IEP developed.
  Arms: Annual Monitoring of IEP
Behavioral: Quarterly Monitoring of IEP — Parents/caregivers and the teacher of participants will be asked to evaluate the effectiveness of the child's IEP four times per academic calendar year. The evaluation is done through the use of an IEP Questionnaire developed for this study. This questionnaire addresses the child's academic performance, progress, and adherence to the IEP developed.
  Arms: Quarterly Monitoring of IEP

SUMMARY:
Neurodevelopmental outcomes in children treated for cancer involving the central nervous system (CNS) provide educators with new challenges with regards to classification, monitoring, and intervention in the regular or special education classroom setting. Recommendations resulting from serial neurodevelopmental evaluations for these children often do not overlap with traditional special education recommendations commonly included in Individual Education Plans (IEPs) for children with congenital or genetic learning problems. The investigators currently do not know whether or not school-based treatment for learning problems, based on the child's IEP, incorporates recommendations made based on a neurodevelopmental evaluation appropriately. In addition, it is not clear whether or not the recommendations that are included in a child's IEP have any beneficial outcome on the child's learning and academic achievement over time. The purpose of this project is to examine the relationship between neurodevelopmental outcomes, recommendations for intervention, special education services and accommodations included in a child's school IEP, and outcome for the child following implementation of the IEP. The study has two major specific aims:

1. To quantify the clinical and educational contributions of recommendations resulting from neurodevelopmental evaluations and the subsequent development of IEPs.

   Hypothesis 1.1: Higher concordance between recommendations made based on neurodevelopmental evaluations and criteria written into children's IEPs will be associated with more positive academic outcomes (i.e. maintenance or improvement in academic skills).

   Hypothesis 1.2: Children who have higher concordance between criteria written into their IEPs and academic services actually received will show more positive academic outcomes than children whose IEP criteria and academic services are less concordant.
2. To evaluate an intervention that will improve academic outcomes for children treated for cancer.

Hypothesis 2.1: Children whose IEPs are monitored more frequently will show more positive academic outcomes than their peers whose IEPs are monitored less frequently.

DETAILED DESCRIPTION:
For years, researchers have examined the effects of cancer and its treatment on children's neurodevelopment. This body of research has identified a number of specific threats to children's cognitive functioning and academic achievement, due to both acute effects and late effects of cancer and its treatment. These often translate into difficulties in the academic setting. Specifically, areas of cognitive and behavioral development are frequently affected, leading to concomitant difficulties in academic achievement and social interaction. Previous research has indicated that such developmental effects and concomitant difficulties are particularly notable in children treated for brain tumors and for leukemias with central nervous system (CNS) involvement. Neurodevelopmental assessments conducted as part of clinical evaluations serve to identify individual strengths and weaknesses of each child treated. Results of these assessments are used to formulate recommendations targeted at compensating for weaknesses by accentuating strengths of each child. Child Study Team meetings are scheduled, at the parent's request, at the child's school in order to use these recommendations in developing Individual Educational Plans (IEPs) to best meet the special needs of the student. At present, no formal follow-up procedure exists to ensure that the IEPs are implemented appropriately, nor that they are effective in meeting the identified special needs of the children.

The present study proposes to 1) evaluate the IEP implementation process for children with cancer, 2) evaluate the effectiveness of IEPs in helping to improve academic outcomes for children with cancer, and 3) to evaluate the influence on academic outcomes of a high-monitoring follow-up intervention for children with cancer. To address these objectives, school-aged children with central nervous system tumors, acute lymphoblastic leukemia, or lymphoma will be administered a neurodevelopmental assessment to measure any specific educational needs they may have. The results of the neurodevelopmental assessment are provided to the parent in a feedback session where any questions or concerns regarding the evaluation can be addressed. At the time of the feedback session, parents are informed of the IEP process and are requested to contact the school to request that a Child Study Team Meeting take place. The study personnel offer to attend the meeting with the parent. Results of the assessments will be used to help guide recommendations made for academic placement and accommodations as per the school's guidelines.

Children with cancer will be assigned to either a quarterly follow-up or annual follow-up group. For those children in the quarterly follow-up group, parents and primary teacher (the primary teacher is identified by the parent/guardian as the teacher who has the most contact with the child and/or knows the child best) will be asked to provide information at the end of each grading period (4 times/year) regarding the child's performance, progress, and adherence to the IEP developed. For children in the yearly follow-up group, this information will only be collected at the end of each academic year. Children in the quarterly and annual follow-up groups will be re-assessed annually for a total of 3 years to evaluate any changes in neurodevelopmental functioning and academic achievement.

Children in the two experimental groups will be administered a neurodevelopmental evaluation, and, in addition, will receive academic follow-up on either a quarterly or annual basis, depending upon to which group they are randomized. Enrollment is on an ongoing basis and each participant will be followed for 3 years after enrollment, receiving a neurodevelopmental evaluation each year with a final endpoint evaluation at year 4 (a total of 4 neurodevelopmental evaluations).

ELIGIBILITY:
Inclusion Criteria:

* Children, ages 6-12 years, who are within 2-5 years of diagnosis for either central nervous system tumor or acute lymphocytic leukemia, or lymphoma at time of enrollment

Exclusion Criteria:

* Children who have been diagnosed with any type of cancer other than a central nervous system tumor, lymphoma, or leukemia.
* Children who are not between the ages of 6-12 years and who were not diagnosed within the past 2-5 years with central nervous system tumor, lymphoma, or leukemia.
* Children who are monolingual in a language other than English or Spanish
* Parent or caregiver of the child is not fluent in English or Spanish
* Child has been diagnosed with a significant mental health disorder that is not responsive to behavioral or medical management. This includes severe depression, schizophrenia, or bipolar disorder. Children whose mental health problem is effectively treated are eligible for participation.

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 62 (Actual)
Dates: Start 2003-01; Primary Completion 2010-10 (Actual); Study Completion 2010-10 (Actual)

PRIMARY OUTCOMES:
Academic achievement as measured by the Woodcock Johnson Tests of Achievement, Third Edition | Measured at Year 1, Year 2 and 3

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Armstrong, PhD, Principal Investigator — University of Miami; Maria L Goldman, PsyD, Study Director — University of Miami
Locations (1):
- Mailman Center for Child Development University of Miami Miller School of Medicine, Miami, Florida, United States